CLINICAL TRIAL: NCT05211466
Title: Digital Care Chains in Health Care - a Study of Care Consumption, Care Quality, Work Environment and Well-being
Status: Completed | Type: Observational
Sponsor: Region Gävleborg (Other)
Collaborators: University of Gavle (Other)
Responsible Party: Sponsor
Other Study IDs: Digital Care Chains
Record Dates: First submitted 2022-01-04; First posted 2022-01-27 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-08

CONDITIONS: Stress and Burnout; Work Environment Adverse Effects; Well-Being, Psychological; Care Givers Satisfaction; Workload; Technology Use
Keywords: Telemedicine; eHealth; Telecare; Telehealth; HIT; care quality; work environment
MeSH Terms: conditions — Burnout, Psychological; Occupational Stress; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Digital care staff: Staff working most of their time (20% or more) with the digital healthcare platform.
  Interventions: Other: Digital healthcare platform
- Traditional care staff: Staff working traditionally, using the digital healthcare platform to a very little extent.

INTERVENTIONS:
Other: Digital healthcare platform — In this specific digital healthcare platform, patients can enter symptoms and get an initial digital triage by artificial intelligence (AI). After the artificial intelligence (AI) has assessed the symptoms, the patient can be triaged to digital healthcare advices, or a chat with a healthcare professional. If needed, the healthcare professional can convert the chat to a telephone or video assessment, or book the patient to a healthcare specialist. The platform can also administer planned consultations with patients or between professionals, it can be used as a tool for the patient to book healthcare appointments, get diagnostics and assessments done, and receive treatment through.
  Groups: Digital care staff

SUMMARY:
Digital healthcare has developed rapidly to meet demands for accessible healthcare, streamline care and meet future challenges with increasing healthcare needs and reduced labour force in Sweden. Developers and stakeholders in Sweden want to exchange the praxis of phone triage to digital or semi-digital triaging tools, to relieve staff's workload and utilize better resource use that would benefit all patient groups. However, previous studies have showed demographic differences in utilization rate and an increase of simpler care matters when digital healthcare options are offered. Also, little is known of medical accuracy of digital triage tools and of the work environment in digital healthcare. More research is needed on this, as well as on care consumption, care quality and of patients' experiences of digital healthcare. The overall aim of the research project is to study a new digital healthcare platform being introduced in 2021/2022 in the County of Gävleborg, Sweden. The studies will focus on care quality and patient safety as well as explore the digital work environment and staff well-being in the digital healthcare platform. Data will be collected before and after the introduction of the digital healthcare platform, using register data and questionnaires. The data from the two time periods will be analyzed with descriptive and inference statistics, to explore if the digital healthcare platform has brought differences on group levels in staff estimates of care quality and patient safety as well as in work environment aspects such as the staffs' well-being.

ELIGIBILITY:
Inclusion Criteria:

* healthcare staff from all clinical areas in the County of Gavleborg
* staff with permanent employment

Exclusion Criteria:

* administrative staff
* managers
* staff on long term leave
* staff on long term sick leave
* staff on parent leave
* staff expected to retire or resign within a year

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be recruited from both public and private healthcare units (amendment of ethical approval number 2021-04696).The study population will consist of professions such as nurses, physicians, physiotherapists and psychologists and will be recruited from in-patient and out-patient care units. 1000-2000 persons will be offered paticipation in each time period.
Sampling Method: Probability Sample
Enrollment: 1012 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2025-01-12 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Staff-reported work environment in digital healthcare compared to traditional healthcare work. | Baseline measure during January - April 2022.
  Questions on work environment will be asked through a survey. The survey contains questions from the following questionnaires: Safety, Communication, Operational Reliability, and Engagement (SCORE) Copenhagen Psychosocial Questionnaire (COPSOQ) Surveys on Patient Safety Culture™ Hospital Survey (SOPS®) and Staff Satisfaction with Care (SSC).
  SCORE: Values between 1-5. Higher scores mean a better outcome in factors on patient safety, working climate and personal growth, with some items reversed. Higher scores mean a worse outcome in factors on workload, burnout and stress.
  COPSOQ: Values between 1-5. Higher scores mean a better outcome in factors on stress and emotional demands, but a worse outcome in factors on workplace community and involvement, with one item reversed.
  SOPS Hospital Survey: Values between 1-5. Higher scores mean a worse outcome. SSC: Values between 1-7. Higher scores mean a better outcome.
Staff-reported well-being in digital healthcare compared to traditional healthcare work. | Baseline measure during January - April 2022.
  Questions on well-being will be asked through a survey. The survey contains questions from the following questionnaires: Safety, Communication, Operational Reliability, and Engagement (SCORE) Copenhagen Psychosocial Questionnaire (COPSOQ) Surveys on Patient Safety Culture™ Hospital Survey (SOPS®) and Staff Satisfaction with Care (SSC).
  SCORE: Values between 1-5. Higher scores mean a better outcome in factors on patient safety, working climate and personal growth, with some items reversed. Higher scores mean a worse outcome in factors on workload, burnout and stress.
  COPSOQ: Values between 1-5. Higher scores mean a better outcome in factors on stress and emotional demands, but a worse outcome in factors on workplace community and involvement, with one item reversed.
  SOPS Hospital Survey: Values between 1-5. Higher scores mean a worse outcome. SSC: Values between 1-7. Higher scores mean a better outcome.
Staff-reported quality of care given through a digital platform compared to traditional healthcare. | Baseline measure during January - April 2022.
  Questions on quality of care will be asked through a survey. The survey contains questions from the following questionnaires: Safety, Communication, Operational Reliability, and Engagement (SCORE) Copenhagen Psychosocial Questionnaire (COPSOQ) Surveys on Patient Safety Culture™ Hospital Survey (SOPS®) and Staff Satisfaction with Care (SSC).
  SCORE: Values between 1-5. Higher scores mean a better outcome in factors on patient safety, working climate and personal growth, with some items reversed. Higher scores mean a worse outcome in factors on workload, burnout and stress.
  COPSOQ: Values between 1-5. Higher scores mean a better outcome in factors on stress and emotional demands, but a worse outcome in factors on workplace community and involvement, with one item reversed.
  SOPS Hospital Survey: Values between 1-5. Higher scores mean a worse outcome. SSC: Values between 1-7. Higher scores mean a better outcome.
Staff-reported work environment in digital healthcare compared to traditional healthcare work. | Measures will be made August to December 2024.
  Questions on work environment will be asked through a survey. The survey contains questions from the following questionnaires: Safety, Communication, Operational Reliability, and Engagement (SCORE) Copenhagen Psychosocial Questionnaire (COPSOQ) Surveys on Patient Safety Culture™ Hospital Survey (SOPS®) and Staff Satisfaction with Care (SSC). Comparisons will be made between time and groups.
  SCORE: Values between 1-5. Higher scores mean a better outcome in factors on patient safety, working climate and personal growth with some items reversed. Higher scores mean a worse outcome in factors on workload, burnout and stress.
  COPSOQ: Values between 1-5. Higher scores mean a better outcome in factors on stress and emotional demands, but a worse outcome in factors on workplace community and involvement with one item reversed.
  SOPS Hospital Survey: Values between 1-5. Higher scores mean a worse outcome. SSC: Values between 1-7. Higher scores mean a better outcome.
Staff-reported well-being in digital healthcare compared to traditional healthcare work. | Measures will be made August to December 2024.
  Questions on well-being will be asked through a survey. The survey contains questions from the following questionnaires: Safety, Communication, Operational Reliability, and Engagement (SCORE) Copenhagen Psychosocial Questionnaire (COPSOQ) Surveys on Patient Safety Culture™ Hospital Survey (SOPS®) and Staff Satisfaction with Care (SSC).
  Comparisons will be made between time and groups. SCORE: Values between 1-5. Higher scores mean a better outcome in factors on patient safety, working climate and personal growth, with some items reversed. Higher scores mean a worse outcome in factors on workload, burnout and stress.
  COPSOQ: Values between 1-5. Higher scores mean a better outcome in factors on stress and emotional demands, but a worse outcome in factors on workplace community and involvement, with one item reversed.
  SOPS Hospital Survey: Values between 1-5. Higher scores mean a worse outcome. SSC: Values between 1-7. Higher scores mean a better outcome.
Staff-reported quality of care given through a digital platform compared to traditional health care. | Measures will be made August to December 2024.
  Questions on quality of care will be asked through a survey. The survey contains questions from the following questionnaires: Safety, Communication, Operational Reliability, and Engagement (SCORE) Copenhagen Psychosocial Questionnaire (COPSOQ) Surveys on Patient Safety Culture™ Hospital Survey (SOPS®) and Staff Satisfaction with Care (SSC).
  Comparisons will be made between time and groups. SCORE: Values between 1-5. Higher scores mean a better outcome in factors on patient safety, working climate and personal growth, with some items reversed. Higher scores mean a worse outcome in factors on workload, burnout and stress.
  COPSOQ: Values between 1-5. Higher scores mean a better outcome in factors on stress and emotional demands, but a worse outcome in factors on workplace community and involvement, with one item reversed.
  SOPS Hospital Survey: Values between 1-5. Higher scores mean a worse outcome. SSC: Values between 1-7. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Agneta C Larsson, MD, PhD, Study Chair — County of Gavleborg
Locations (1):
- County of Gavleborg, Gävle, Gävleborg County, Sweden

IPD SHARING:
Plan to Share IPD: No
Due to the General Data Protection Regulation (GDPR) and restrictions in ethical approvement, individual data can not be shared. Protocols and statistics not including individual data, can be shared eventually. Informed consent forms can be shared.

REFERENCES:
- [Background] Ekman B, Thulesius H, Wilkens J, Lindgren A, Cronberg O, Arvidsson E. Utilization of digital primary care in Sweden: Descriptive analysis of claims data on demographics, socioeconomics, and diagnoses. Int J Med Inform. 2019 Jul;127:134-140. doi: 10.1016/j.ijmedinf.2019.04.016. Epub 2019 Apr 22. PMID 31128825
- [Background] Gabrielsson-Jarhult F, Kjellstrom S, Josefsson KA. Telemedicine consultations with physicians in Swedish primary care: a mixed methods study of users' experiences and care patterns. Scand J Prim Health Care. 2021 Jun;39(2):204-213. doi: 10.1080/02813432.2021.1913904. Epub 2021 May 11. PMID 33974502
- [Background] Ashwood JS, Mehrotra A, Cowling D, Uscher-Pines L. Direct-To-Consumer Telehealth May Increase Access To Care But Does Not Decrease Spending. Health Aff (Millwood). 2017 Mar 1;36(3):485-491. doi: 10.1377/hlthaff.2016.1130. PMID 28264950
- [Background] Shah SJ, Schwamm LH, Cohen AB, Simoni MR, Estrada J, Matiello M, Venkataramani A, Rao SK. Virtual Visits Partially Replaced In-Person Visits In An ACO-Based Medical Specialty Practice. Health Aff (Millwood). 2018 Dec;37(12):2045-2051. doi: 10.1377/hlthaff.2018.05105. PMID 30633681
- [Background] Totten AM, Womack DM, Eden KB, McDonagh MS, Griffin JC, Grusing S, Hersh WR. Telehealth: Mapping the Evidence for Patient Outcomes From Systematic Reviews [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2016 Jun. Report No.: 16-EHC034-EF. Available from http://www.ncbi.nlm.nih.gov/books/NBK379320/ PMID 27536752
- [Background] Fraser H, Coiera E, Wong D. Safety of patient-facing digital symptom checkers. Lancet. 2018 Nov 24;392(10161):2263-2264. doi: 10.1016/S0140-6736(18)32819-8. Epub 2018 Nov 6. No abstract available. PMID 30413281
- [Background] Kroth PJ, Morioka-Douglas N, Veres S, Babbott S, Poplau S, Qeadan F, Parshall C, Corrigan K, Linzer M. Association of Electronic Health Record Design and Use Factors With Clinician Stress and Burnout. JAMA Netw Open. 2019 Aug 2;2(8):e199609. doi: 10.1001/jamanetworkopen.2019.9609. PMID 31418810
- [Background] Alami H, Gagnon MP, Fortin JP. Some Multidimensional Unintended Consequences of Telehealth Utilization: A Multi-Project Evaluation Synthesis. Int J Health Policy Manag. 2019 Jun 1;8(6):337-352. doi: 10.15171/ijhpm.2019.12. PMID 31256566